CLINICAL TRIAL: NCT06722417
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Icalcaprant in Healthy Adult Japanese and Han Chinese Subjects
Brief Title: A Single Dose Study to Assess Adverse Events and How Oral Icalcaprant Moves Through the Body in Healthy Adult Japanese and Han Chinese Participants
Acronym: 528 Asian PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M25-528
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Icalcaprant; ABBV-1354; CVL-354

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Icalcaprant Dose A- Japanese Participants (Experimental): Participants will receive oral Icalcaprant dose A once, then a 30-day follow-up period.
  Interventions: Drug: Icalcaprant
- Group 2: Icalcaprant Dose A- Han Chinese Participants (Experimental): Participants will receive oral Icalcaprant dose A once, then a 30-day follow-up period.
  Interventions: Drug: Icalcaprant

INTERVENTIONS:
Drug: Icalcaprant — Oral capsules
  Other Names: ABBV-1354; CVL-354

SUMMARY:
This study will assess the pharmacokinetics, safety, and tolerability of icalcaprant administered orally in healthy adult Japanese and Han Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese or Han Chinese individuals.
* Japanese participants must be first or second-generation Japanese of full Japanese parentage. First-generation participants will have been born in Japan to two parents and four grandparents also born in Japan of full Japanese descent. Second-generation participants born outside of Japan must have two parents and four grandparents born in Japan of full Japanese descent. All participants must maintain a typical Japanese lifestyle, including consuming a typical Japanese diet.
* Han Chinese participants must be first or second-generation Han Chinese of full Chinese parentage. First-generation participants will have been born in China to two parents and four grandparents also born in China of full Han Chinese descent. Second-generation participants born outside of China must have two parents and four grandparents born in China of full Han Chinese descent. Participants must maintain a typical Chinese lifestyle, including consuming a typical Chinese diet.
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of epilepsy, seizure (except febrile seizure during childhood), unexplained alteration of consciousness, head injury with associated loss of consciousness, sleep disorder (except mild insomnia not requiring daily therapy), any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness. - History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.
* No use of tobacco or nicotine-containing products within 180 days prior to the first dose of study drug.
* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Icalcaprant | Up to approximately 6 days
  Cmax of Icalcaprant
Time to Cmax (Tmax) of Icalcaprant | Up to approximately 6 days
  Tmax of Icalcaprant
Terminal Phase Elimination Rate Constant (Beta) of Icalcaprant | Up to approximately 6 days
  Beta of Icalcaprant
Terminal Phase Elimination Half-Life (t1/2) of Icalcaprant | Up to approximately 6 days
  T1/2 of Icalcaprant
Area under the plasma concentration-time curve from time 0 until the last measurable Concentration (AUCt) of Icalcaprant | Up to approximately 6 days
  AUCt of Icalcaprant
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of Icalcaprant | Up to approximately 6 days
  AUCinf of Icalcaprant
Number of Participants with Adverse Events (AEs) | Up to approximately 37 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Anaheim Clinical Trials, LLC /ID# 271323, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-528